CLINICAL TRIAL: NCT06084130
Title: The Effect of Zolpidem on CPAP Acclimatization in Patients With OSA: A Crossover, Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Zolpidem on CPAP Acclimatization in OSA
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Navarat Kasemsuk, Clinical Educator, Siriraj Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 365/2566[IRB4]
Record Dates: First submitted 2023-09-28; First posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Zolpidem

STUDY DESIGN:
Intervention Model Description: The eligible participants will be informed and consented. After then, the participants in group 1 will receive 10 milligrams zolpidem contained in white-color opaque medicine capsule prepared by the pharmacist, meanwhile the participants in group 2 will receive placebo which is corn-starch contained in identical white-color opaque medicine capsule. The participants will be advised to take the medication 30 minutes prior to the bedtime until the 1-week follow up visit. On the second week, the participants in group 1 will alternatively receive placebo, meanwhile the participants in group 2 will receive 10 milligrams zolpidem in identical capsules. The wash-out period is 24 hours as the fact that the half-life of zolpidem is 2 hours and total zolpidem elimination time is 10 to 12 hours.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebo is corn-starch contained in identical white-color opaque medicine capsule to zolpidem
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zolpidem (Experimental): The participants in Zolpidem group will receive 10 milligrams zolpidem contained in white-color opaque medicine capsule prepared by the pharmacist. The participants will be advised to take the medication 30 minutes prior to the bedtime until the 1-week follow up visit.
  Interventions: Drug: Zolpidem
- Placebo (Placebo Comparator): The participants in Placebo group will receive placebo which is corn-starch contained in identical white-color opaque medicine capsule. The participants will be advised to take the medication 30 minutes prior to the bedtime until the 1-week follow up visit.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zolpidem — 10 milligrams zolpidem contained in white-color opaque medicine capsule
  Arms: Zolpidem
Drug: Placebo — corn-starch contained in identical white-color opaque medicine capsule
  Arms: Placebo

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder characterized by a cessation or significant decrease in airflow during sleep. CPAP is the preferred therapy and has high effectiveness at all levels of OSA severity. It acts as a pneumatic splint to maintain upper airway patency during sleep, preventing the soft tissues from collapsing. However, the patient's compliance continues to be an issue. One of the main contributors to CPAP therapy failure is difficulty falling asleep. To aid in the machine's adaptation, hypnotic medicine was administered.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a sleep disorder characterized by a cessation or significant decrease in airflow during sleep. According to a recent study, OSA may impact over 1 billion individuals worldwide. In Thailand, the prevalence of snoring in children is 6.9-8.5%, while the prevalence of OSA in children is 0.7-1.3%. Moreover, OSA affects 15.4% of Thai male adults and 6.3% of Thai females. Untreated OSA can lead to daytime sleepiness, decreased productivity, increased motor vehicle accidents, and worsening hypertension, atrial fibrillation, and stroke. Oral appliances, upper airway surgery, and continuous positive airway pressure (CPAP) devices are available as treatment alternatives.

CPAP is the preferred therapy and has high effectiveness at all levels of OSA severity. It acts as a pneumatic splint to maintain upper airway patency during sleep, preventing the soft tissues from collapsing. Through this mechanism, it effectively eliminates the apneas and/or hypopneas, decreases the arousals, and normalizes the oxygen saturation. However, the patient's compliance continues to be an issue. Failure of CPAP therapy may occur in up to 25% to 50% of patients, with patients typically discontinuing therapy within the first 2 to 4 weeks of treatment and 91% of patients discontinuing CPAP therapy within the first three years of therapy.

According to the clinical guidelines of the American Academy of Sleep Medicine, all potential PAP titration candidates should receive adequate PAP education, hands-on demonstration, careful mask fitting, and acclimatization prior to titration. Acclimatization is a technique used to familiarize patients with PAP therapy for compliance.

One of the main contributors to CPAP therapy failure is difficulty falling asleep. To aid in the machine's adaptation, hypnotic medicine was administered. Sedative medications now came in a variety of categories. Non-benzodiazepines sometimes referred to as Z-drugs, are among those with the beneficial characteristics of not deteriorating OSA severity, not contributing to drug addiction, possessing a rapid onset, and exhibiting fewer adverse consequences. Zolpidem, eszopiclone and zaleplon are included in this drug class. According to a previous meta-analysis, eszopiclone greatly facilitated the use of CPAP. However, up until now limited research on zolpidem and zaleplon was conducted. This study aims to evaluate the effect of zolpidem on CPAP compliance in OSA patients as compared to a placebo.

ELIGIBILITY:
Inclusion Criteria:

* OSA patients whose sleep test demonstrated apnea-hypopnea index (AHI) ≥ 15 /hour or AHI ≥ 5 /hour with comorbid disease including hypertension, cardiovascular disease, and stroke
* Age 18 to 75 years
* Indicated for CPAP therapy
* Naïve for the device usage

Exclusion Criteria:

* A history of zolpidem allergies
* Currently take hypnotic medications
* Denied permission to engage in the study and/or follow its protocol
* Individuals with liver diseases, including hepatitis from any cause, liver cirrhosis, and liver cancer

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-15 (Estimated); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
CPAP hour usage per night | on the end of the 1st as the 1st follow-up and the 2nd week as the 2nd follow-up
  CPAP hour usage per night in hours

SECONDARY OUTCOMES:
Numbers of the patients with CPAP usage ≥ 4 hours | on the end of the 1st as the 1st follow-up and the 2nd week as the 2nd follow-up
  Numbers of the patients with CPAP usage ≥ 4 hours in persons
Number of the participants with % CPAP usage ≥ 70 | on the end of the 1st as the 1st follow-up and the 2nd week as the 2nd follow-up
  Number of the participants with % CPAP usage ≥ 70 in persons
drug compliance, and adverse events | on the end of the 1st as the 1st follow-up and the 2nd week as the 2nd follow-up
  drug compliance with residual drug counts, and adverse events reports

REFERENCES:
- [Derived] Pisalnoradej P, Banhiran W, Kasemsuk N. The effect of zolpidem on CPAP acclimatization in patients with OSA: a crossover, randomized, double-blinded, placebo-controlled trial. J Clin Sleep Med. 2025 Nov 1;21(11):1831-1837. doi: 10.5664/jcsm.11850. PMID 40790926

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT06084130/Prot_SAP_000.pdf
  • Informed Consent Form (2023-10-09): https://cdn.clinicaltrials.gov/large-docs/30/NCT06084130/ICF_001.pdf